CLINICAL TRIAL: NCT02255591
Title: Shamrock Versus Lumbar Ultrasound Trident - Ultrasound Guided Block of the Lumbar Plexus: A Randomized Controlled Trial
Brief Title: Shamrock Versus Lumbar Ultrasound Trident - Ultrasound Guided Block of the Lumbar Plexus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: AP Moeller Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AUH-TFB-SR; 2013-005346-10 (EudraCT Number)
Record Dates: First submitted 2014-09-22; First posted 2014-10-02 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2014-09

CONDITIONS: Hip Fractures; Anesthesia Local; Pain, Postoperative
Keywords: Hip surgery anesthesia; Perioperative analgesia
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shamrock (Experimental): Use of the Shamrock technique to place a lumbar plexus block with injection of 20 mL 2% Lidocaine-adrenaline added gadolinium.
  Interventions: Drug: Lidocaine-adrenaline added gadolinium.
- Lumbar Ultrasound Trident (Active Comparator): Use of the Lumbar Ultrasound Trident technique to place a lumbar plexus block with injection of 20 mL 2% lidocaine-adrenaline added gadolinium.
  Interventions: Drug: Lidocaine-adrenaline added gadolinium.

INTERVENTIONS:
Drug: Lidocaine-adrenaline added gadolinium.

SUMMARY:
The main objective of the trial is to complete a double-blinded randomized controlled trial of a lumbar plexus block with the Shamrock technique versus the Lumbar Ultrasound Trident technique by estimating the time of performance of lumbar plexus blocks in healthy volunteers.

Secondary objectives include a) estimates of number and depth of needle injections, distance of injection site from the midline, minimal electric nerve stimulation to trigger muscular response and the type of response, and volunteer discomfort during block injection, b) measurements of plasma lidocaine and mean arterial blood pressure, c) examinations of sensory block of the dermatomes T8-S3 and motor block of the femoral nerve, the obturator nerve, the hip abductor muscles, and the hamstring muscles, d) success rate of lumbar plexus block, e) perineural and epidural distribution of local anesthetics added contrast visualized on magnetic resonance imaging (MRI) scanning, and f) cost-effectiveness for the Shamrock technique versus the Lumbar Ultrasound Trident Technique for lumbar plexus block in healthy volunteers.

The hypothesis is that the Shamrock technique is faster to perform than the Lumbar Ultrasound technique, and that the success rate of the Shamrock technique is equal to or higher than the Lumbar Ultrasound Trident technique.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥ 18 years
* Volunteers who have given their written and oral consent to participate in the study after fully understanding the content and the limitations of the protocol
* Normal healthy volunteer (American Society of Anesthesiology (ASA) Classification I)

Exclusion Criteria:

* Volunteers not able to cooperate for the study
* Volunteers not able to understand Danish
* Daily use of analgesics
* Allergy against the medicines used in the study
* Drug abuse (according to the investigator's judgement)
* Alcohol consumption larger than the recommendations of the Danish National Board of Health
* Volunteers in whom nerve blocks are not possible due to technical reasons
* Volunteers who meet any contraindication for MRI including claustrophobia
* Volunteers who are incompetent, i.e. surrogate consent is not accepted

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Block performance time | Estimated 0 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Time for performance of lumbar plexus block in seconds from placement of the ultrasound transducer on the skin until the block needle is pulled out after injection of local anesthetics.

SECONDARY OUTCOMES:
Number of needle feeds | Estimated 0 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Needle feeds are defined as retraction of needle followed by new feed of the needle disregarding the number of skin punctures.
Discomfort during block placement | Estimated 1 minute after block placement. Presented 10 months after the last visit of the last volunteer.
  Discomfort is measured with Numeric Rating Scale (NRS).
Plasma Lidocaine | Blood samples are withdrawn 0, 5, 10, 20, 40, 60, and 90 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
Mear arterial pressure | Measured 5 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
Cost-effectiveness | Calculated two weeks after the last visit of the last volunteer. Presented 10 months after the last visit of the last volunteer.
  Cost-effectiveness estimated as extra expense per successful lumbar plexus block and calculated as incremental cost-effectiveness ratio (ICER).
Sensor block | Tested 30 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Sensor block (cold, warm, touch, and pain) of the dermatomes T8-S3 and of the femoral nerve and the lateral femoral cutaneous nerve.
Motor block | Tested 40 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Motor block of the femoral nerve (knee extension), the obturator nerve (hip adduction), the superior gluteal nerve (hip abduction), and the sciatic nerve (knee flexion) estimated as active resistance against movement of the relevant joint and with sphygmomanometer of the relevant joint as maximal voluntary isometric contraction with dynamometer (mmHg).
Block success rate | Tested 30 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Success rate defined as motor block of the femoral nerve (knee extension) and the obturator nerve (hip adduction) and reduced sensory of the lateral femoral cutaneous nerve (middle of the lateral side of the thigh).
Block success rate | Tested 30 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Defined as above after lumbar plexus block with the Shamrock technique for motor response on electrical nerve stimulation above respectively below 0,5 milliampere (mA).
Epidural spread of local anesthetics with contrast | Estimated 10-30 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Estimated with T1- and T2-weighted and with diffusion weighted imaging (DWI) MR scanning.
Perineural spread of local anesthetics with added contrast | Estimated 10-30 minutes after block placement. Presented 10 months after the last visit of the last volunteer.
  Estimated with T1- and T2-weighted and with DWI MR scanning.
Depth of block needle | Estimated during block
  The depth in cm from the injection site in the skin to the needle tips position during injection. of local anesthetics
Injection site | Estimated immediately after block placement
  The distance in cm from the injection site of the block needle to the midline of the volunteer.
Minimal electrical nerve stimulation | Estimated immediately before injection of local anesthetics during block placement
  The estimated minimal electrical nerve stimulation in mA to trigger a muscular response.
Type of response on electrical nerve stimulation | Assessed immediately before injection of local anesthetics during block placement
  The type of response triggered by electrical nerve stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Bendtsen, MD,PhD,Prof., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Aarhus University Hospital, Noerrebrogade 44, DK-8000 Aarhus C, Denmark
Locations (1):
- Department of Aneshtesiology and Intensive Care Medicine; Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] de Visme V, Picart F, Le Jouan R, Legrand A, Savry C, Morin V. Combined lumbar and sacral plexus block compared with plain bupivacaine spinal anesthesia for hip fractures in the elderly. Reg Anesth Pain Med. 2000 Mar-Apr;25(2):158-62. doi: 10.1053/rapm.2000.0250158. PMID 10746528
- [Background] Kirchmair L, Entner T, Kapral S, Mitterschiffthaler G. Ultrasound guidance for the psoas compartment block: an imaging study. Anesth Analg. 2002 Mar;94(3):706-10; table of contents. doi: 10.1097/00000539-200203000-00042. PMID 11867402
- [Background] Kirchmair L, Entner T, Wissel J, Moriggl B, Kapral S, Mitterschiffthaler G. A study of the paravertebral anatomy for ultrasound-guided posterior lumbar plexus block. Anesth Analg. 2001 Aug;93(2):477-81, 4th contents page. doi: 10.1097/00000539-200108000-00047. PMID 11473883
- [Background] Morimoto M, Kim JT, Popovic J, Jain S, Bekker A. Ultrasound-guided lumbar plexus block for open reduction and internal fixation of hip fracture. Pain Pract. 2006 Jun;6(2):124-6. doi: 10.1111/j.1533-2500.2006.00074.x. PMID 17309721
- [Background] Doi K, Sakura S, Hara K. A modified posterior approach to lumbar plexus block using a transverse ultrasound image and an approach from the lateral border of the transducer. Anaesth Intensive Care. 2010 Jan;38(1):213-4. No abstract available. PMID 20191806
- [Background] Madison SJ, Ilfeld BM, Loland VJ, Mariano ER. Posterior lumbar plexus perineural catheter insertion by ultrasound guidance alone. Acta Anaesthesiol Scand. 2011 Sep;55(8):1031-2. doi: 10.1111/j.1399-6576.2011.02489.x. Epub 2011 Jul 20. No abstract available. PMID 21770905
- [Background] Karmakar MK, Ho AM, Li X, Kwok WH, Tsang K, Ngan Kee WD. Ultrasound-guided lumbar plexus block through the acoustic window of the lumbar ultrasound trident. Br J Anaesth. 2008 Apr;100(4):533-7. doi: 10.1093/bja/aen026. PMID 18344573
- [Derived] Strid JMC, Sauter AR, Ullensvang K, Andersen MN, Daugaard M, Bendtsen MAF, Soballe K, Pedersen EM, Borglum J, Bendtsen TF. Ultrasound-guided lumbar plexus block in volunteers; a randomized controlled trial. Br J Anaesth. 2017 Mar 1;118(3):430-438. doi: 10.1093/bja/aew464. PMID 28203808